CLINICAL TRIAL: NCT00141310
Title: A Randomised, Double-Blind, Placebo-Controlled, Flexible-Dose, Parallel-Group Study to Evaluate the Efficacy, Safety and Toleration of Oral Sildenafil Citrate Administered in the Dose Range of 20 - 80 Mg TID for the Treatment of Pre-Eclampsia. (PET)
Brief Title: Sildenafil Citrate for the Treatment of Established Pre-Eclampsia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study prematurely discont'd 20-Apr-2006 after interim analysis suggested sample size could be reduced without losing power. No safety concerns led to decision.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1481206
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Pre-eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: Sildenafil citrate

SUMMARY:
To determine the efficacy and safety of sildenafil citrate in the treatment of established pre-eclampsia

ELIGIBILITY:
Inclusion Criteria:

* Subjects with pre-eclampsia defined as new hypertension with a diastolic BP of > or = 90 mmHg on two occasions separated by at least 4 hrs arising after 20 weeks of pregnancy, associated with >500 mg/24 hr proteinuria. Subjects with pre-existing hypertension (on treatment) need only fulfill proteinuria requirement.
* Gestational age 24-34 w
* Singleton pregnancy

Exclusion Criteria:

* Where urgent delivery is indicated
* Where the fetus is suspected to have a structural or chromosomal abnormality

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76
Dates: Start 2004-09; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Primary endpoint is the time from randomization to delivery.

SECONDARY OUTCOMES:
Individualised birth-weight ratio at delivery, Placental weight, Umbilical artery pulsatility index, Other indices of PET (incl. uric acid and maternal BP), Safety and toleration, Population PK, Fetal exposure (PK)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United Kingdom (8):
  - Pfizer Investigational Site, Pembury, Kent
  - Pfizer Investigational Site, Royal Tunbridge Wells, Kent
  - Pfizer Investigational Site, Ashton-under-Lyne, Lancs
  - Pfizer Investigational Site, Bolton
  - Pfizer Investigational Site, Dundee
  - Pfizer Investigational Site, Fife
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Manchester

REFERENCES:
- [Derived] Samangaya RA, Mires G, Shennan A, Skillern L, Howe D, McLeod A, Baker PN. A randomised, double-blinded, placebo-controlled study of the phosphodiesterase type 5 inhibitor sildenafil for the treatment of preeclampsia. Hypertens Pregnancy. 2009 Aug;28(4):369-82. doi: 10.3109/10641950802601278. PMID 19843000
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481206&StudyName=Sildenafil%20Citrate%20for%20the%20Treatment%20of%20Established%20Pre-Eclampsia